CLINICAL TRIAL: NCT00882661
Title: A Prospective Randomized Clinical Investigation of the SECURE-C Cervical Artificial Disc: A Pivotal Study/ SECURE-C Cervical Artificial Disc Postmarket Approval Study
Brief Title: SECURE®-C Cervical Artificial Disc Clinical Study/ SECURE-C Cervical Artificial Disc Postmarket Approval Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Globus Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GPR002
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Symptomatic Cervical Disc Disease
Keywords: Neck Pain; Arm Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- SECURE-C Cervical Artificial Disc (Experimental): Treatment of symptomatic cervical disc disease with the SECURE-C Cervical Artificial Disc
  Interventions: Device: SECURE-C Cervical Artificial Disc
- ASSURE Cervical plate and an allograft interbody spacer (Active Comparator): Treatment of symptomatic cervical disc disease utilizing an instrumented anterior discectomy and interbody fusion
  Interventions: Device: ASSURE Cervical plate and an allograft interbody spacer

INTERVENTIONS:
Device: SECURE-C Cervical Artificial Disc — Treatment of symptomatic cervical disc disease with the SECURE-C Cervical Artificial Disc
  Arms: SECURE-C Cervical Artificial Disc
Device: ASSURE Cervical plate and an allograft interbody spacer — Treatment of symptomatic cervical disc disease utilizing an instrumented anterior discectomy and interbody fusion
  Arms: ASSURE Cervical plate and an allograft interbody spacer

SUMMARY:
The purpose of the pivotal IDE clinical study was to evaluate the safety and effectiveness of the SECURE®-C Cervical Artificial Disc for the treatment of symptomatic cervical disc disease at one level between C3 and C7, compared to anterior cervical discectomy and fusion.

The purpose of the Postmarket Approval Study is to evaluate the long-term safety and efficacy associated with the use of the SECURE-C Cervical Artificial Disc

DETAILED DESCRIPTION:
Ages Eligible for Study: 18 to 60 years

Genders Eligible for Study: Both

Accepts Healthy Volunteers: No

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic cervical disc disease (SCDD) in one vertebral level between C3-C7, defined as neck or arm (radicular) pain, or functional or neurological deficit and radiographic confirmation (by CT, MRI, X-ray, etc.) of any of the following:
* Herniated nucleus pulposus;
* Radiculopathy or myelopathy;
* Spondylosis (defined by the presence of osteophytes); or
* Loss of disc height.
* Age between 18 and 60 years
* Failed at least 6 weeks of conservative treatment
* Neck Disability Index (NDI) Questionnaire score of at least 30 (as percentage of 50 point total)
* Able to understand and sign informed consent form
* Psychosocially, mentally and physically able to fully comply with this protocol including adhering to follow-up schedule and filling out forms
* Able to meet the proposed follow-up schedule at 6 weeks, 3 months, 6 months, 12 months and 24 months
* Able to follow postoperative management program

Exclusion Criteria:

* More than one vertebral level requiring treatment
* Prior fusion surgery adjacent to the vertebral level being treated
* Prior surgery at the level to be treated
* Clinically compromised vertebral bodies at the affected level(s) due to current or past trauma
* Radiographic confirmation of facet joint disease or degeneration, defined as apparent sclerosis and/or hypertrophy of the facets demonstrated on AP radiographs as a disruption of the normally smooth facet curve
* Marked cervical instability on resting lateral or flexion/extension radiographs:
* Translation greater than 3mm, and/or
* More than 11° of rotational difference from that of either adjacent level.
* Severe spondylosis at the level to be treated as characterized by any of the following:
* Bridging osteophytes;
* A loss of disc height greater than 50%; or
* Absence of motion (<2°)
* Neck or arm pain of unknown etiology
* Osteoporosis, osteopenia, Paget's disease, osteomalacia or any other metabolic bone disease
* Pregnant or interested in becoming pregnant in the next 2 years
* Active systemic or local infection
* Known allergy to titanium, polyethylene, cobalt, chromium or molybdenum
* Taking medications or any drug known to potentially interfere with bone/soft tissue healing (e.g., steroids)
* Rheumatoid arthritis or other autoimmune disease
* Systemic disease including AIDS, HIV, Hepatitis
* Active malignancy: A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless he/she has been treated with curative intent and there has been no clinical signs or symptoms of the malignancy for at least 5 years
* Neuromuscular disorders such as muscular dystrophy, spinal muscular atrophy, amyotrophic lateral sclerosis, etc.
* Acute mental illness or substance abuse
* Use of bone growth stimulator within past 30 days
* Participation in other investigational device or drug clinical trials within 30 days of surgery
* Prisoners

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 380 (Actual)
Dates: Start 2005-07; Primary Completion 2010-04 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Marzluff, MD, Principal Investigator — Trident Regional Medical Center

RESULTS

PARTICIPANT FLOW:
Period: Investigational Training
Arm/Group | SECURE-C Cervical Artificial Disc | ASSURE Cervical Plate and an Allograft Interbody Spacer
Started | 89 | 0
Completed | 79 | 0
Not Completed | 10 | 0
Period: Treatment
Arm/Group | SECURE-C Cervical Artificial Disc | ASSURE Cervical Plate and an Allograft Interbody Spacer
Started | 151 | 140
Completed | 141 | 114
Not Completed | 10 | 26

BASELINE CHARACTERISTICS:
Groups:
- Randomized SECURE-C Cervical Artificial Disc: Treatment of symptomatic cervical disc disease with the SECURE-C Cervical Artificial Disc
- ASSURE Cervical Plate and Allograft Interbody Spacer: Treatment of symptomatic cervical disc disease utilizing an instrumented anterior discectomy and interbody fusion
- Non-Randomized SECURE-C Cervical Artificial Disc: The first five subjects enrolled at each center were non-randomized subjects receiving the SECURE-C Cervical Artificial Disc
- Total: Total of all reporting groups
Arm/Group | Randomized SECURE-C Cervical Artificial Disc | ASSURE Cervical Plate and Allograft Interbody Spacer | Non-Randomized SECURE-C Cervical Artificial Disc | Total
Number analyzed (Participants) | 151 | 140 | 89 | 380
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (7.5) | 44.4 (7.9) | 41.6 (8.13) | 43.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 72 | 42 | 184
  Male | 81 | 68 | 47 | 196
Region of Enrollment [Number; unit: participants]
  United States | 151 | 140 | 89 | 291

OUTCOME MEASURES:

1. Primary Outcome: Individual Patient Overall Success
Description: Individual patient overall success defined as pain/disability improvement of at least 25% in Neck Disability Index (NDI) compared to baseline; no device failures requiring revision, removal, reoperation, or supplemental fixation; absence of major complications defined as major vessel injury, neurological damage, or nerve injury; and for control fusion patients only, radiographic fusion
Time Frame: 24 months
Population: At the time of database lock, of the 380 patients enrolled in the PMA study, all had reached the 24 month post-operative visit. Complete primary endpoint data was available for 79 Non-randomized SECURE-C patients,141 randomized SECURE-C patients and 114 control patients at 24 months.
Measure: Number; unit: participants
Arm/Group | Randomized SECURE-C Cervical Artificial Disc | ASSURE Cervical Plate and an Allograft Interbody Spacer | Non-Randomized SECURE-C Cervical Artificial Disc
Number analyzed (Participants) | 141 | 114 | 79
participants | 127 | 81 | 67

2. Secondary Outcome: Neck Disability Index (NDI)
Description: Neck Disability Index (NDI) success defined as ≥25% improvement at 24 months from baseline
Time Frame: 24 months
Population: At the time of database lock, of the 380 patients enrolled in the PMA study, all had reached the 24 month post-operative visit. Complete Neck Disability Index (NDI) data was available for 78 Non-randomized SECURE-C patients,139 randomized SECURE-C patients and 116 control patients at 24 months.
Measure: Number; unit: participants
Arm/Group | Randomized SECURE-C Cervical Artificial Disc | ASSURE Cervical Plate and an Allograft Interbody Spacer | Non-Randomized SECURE-C Cervical Artificial Disc
Number analyzed (Participants) | 139 | 116 | 78
participants | 127 | 101 | 67

3. Secondary Outcome: Neck Pain Visual Analog Scale (VAS)
Description: Improvement of 20mm from baseline in neck pain measured using the Visual Analog Scale (VAS)
Time Frame: 24 months
Population: At the time of database lock, of the 380 patients enrolled in the PMA study, all had reached the 24 month post-operative visit. Complete Neck Pain Visual Analog Scale (VAS) data was available for 75 non-randomized SECURE-C, 133 randomized SECURE-C patients and 108 control patients at 24 months.
Measure: Number; unit: participants
Arm/Group | Randomized SECURE-C Cervical Artificial Disc | ASSURE Cervical Plate and an Allograft Interbody Spacer | Non-Randomized SECURE-C Cervical Artificial Disc
Number analyzed (Participants) | 133 | 108 | 75
participants | 104 | 76 | 54

4. Secondary Outcome: Left Arm Pain Visual Analog Scale (VAS)
Description: Improvement of 20mm from baseline in left arm pain measured using the Visual Analog Scale (VAS)
Time Frame: 24 months
Population: At the time of database lock, of the 380 patients enrolled in the PMA study, all had reached the 24 month post-operative visit. Complete Left Arm Pain Visual Analog Scale (VAS) data was available for 75 non-randomized SECURE-C, 133 randomized SECURE-C patients and 108 control patients at 24 months.
Measure: Number; unit: participants
Arm/Group | Randomized SECURE-C Cervical Artificial Disc | ASSURE Cervical Plate and an Allograft Interbody Spacer | Non-Randomized SECURE-C Cervical Artificial Disc
Number analyzed (Participants) | 133 | 108 | 75
participants | 74 | 55 | 37

5. Secondary Outcome: Right Arm Pain Visual Analog Scale (VAS)
Description: Improvement of 20mm from baseline in right arm pain measured using the Visual Analog Scale (VAS)
Time Frame: 24 months
Population: At the time of database lock, of the 380 patients enrolled in the PMA study, all had reached the 24 month post-operative visit. Complete Right Arm Pain Visual Analog Scale (VAS) data was available for 75 non-randomized SECURE-C patients, 133 randomized SECURE-C patients and 108 control patients at 24 months.
Measure: Number; unit: participants
Arm/Group | Randomized SECURE-C Cervical Artificial Disc | ASSURE Cervical Plate and an Allograft Interbody Spacer | Non-Randomized SECURE-C Cervical Artificial Disc
Number analyzed (Participants) | 133 | 108 | 75
participants | 57 | 49 | 36

6. Secondary Outcome: SF-36 PCS
Description: Health Status Survey SF-36 physical composite scores: 15% improvement from baseline
Time Frame: 24 months
Population: At the time of database lock, of the 380 patients enrolled in the PMA study, all had reached the 24 month post-operative visit. Complete SF-36 PCS data was available for 78 non-randomized SECURE-C patients, 138 randomized SECURE-C patients and 114 control patients at 24 months.
Measure: Number; unit: participants
Arm/Group | Randomized SECURE-C Cervical Artificial Disc | ASSURE Cervical Plate and an Allograft Interbody Spacer | Non-Randomized SECURE-C Cervical Artificial Disc
Number analyzed (Participants) | 138 | 114 | 78
participants | 109 | 89 | 53

7. Secondary Outcome: SF-36 MCS
Description: Health Status Survey SF-36 mental composite scores: 15% improvement from baseline
Time Frame: 24 months
Population: At the time of database lock, of the 380 patients enrolled in the PMA study, all had reached the 24 month post-operative visit. Complete SF-36 MCS data was available for 78 non-randomized SECURE-C patients, 138 randomized SECURE-C patients and 114 control patients at 24 months.
Measure: Number; unit: participants
Arm/Group | Randomized SECURE-C Cervical Artificial Disc | ASSURE Cervical Plate and an Allograft Interbody Spacer | Non-Randomized SECURE-C Cervical Artificial Disc
Number analyzed (Participants) | 138 | 114 | 78
participants | 70 | 48 | 45

8. Secondary Outcome: Satisfaction
Description: Patient satisfaction (definitely/mostly): proportion of patients
Time Frame: 24 months
Population: At the time of database lock, of the 380 patients enrolled in the PMA study, all had reached the 24 month post-operative visit. Complete Patient Satisfaction data was available for 78 non-randomized SECURE-C patients, 139 randomized SECURE-C patients and 115 control patients at 24 months.
Measure: Number; unit: participants
Arm/Group | Randomized SECURE-C Cervical Artificial Disc | ASSURE Cervical Plate and an Allograft Interbody Spacer | Non-Randomized SECURE-C Cervical Artificial Disc
Number analyzed (Participants) | 139 | 115 | 78
participants | 133 | 98 | 72

ADVERSE EVENTS:
Time Frame: 24 months
Description: The analysis of safety was based on the as-treated cohort of 380 total patients (88 non-randomized SECURE-C patients, 148 randomized SECURE-C patients, and 144 ACDF patients). The control ACDF group includes 140 patients randomized to ACDF, 3 patients randomized to SECURE-C who received ACDF, and 1 patient from the non-randomized cohort who received ACDF. The Clinical Events Committee (CEC) classified each adverse event.
Arm/Group | SECURE-C Cervical Artificial Disc | ASSURE Cervical Plate and an Allograft Interbody Spacer
Serious Adverse Events (participants affected / at risk) | 46/236 | 34/144
Other Adverse Events (participants affected / at risk) | 121/236 | 80/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SECURE-C Cervical Artificial Disc (N=236) | ASSURE Cervical Plate and an Allograft Interbody Spacer (N=144)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cardiovascular (Cardiac disorders) | 5 | 0
Carpal Tunnel Syndrome (CTS) (General disorders) | 6 | 3
Cerebrovascular (Vascular disorders) | 2 | 0
Compressive Periph Neuro (Non-CTS) (Nervous system disorders) | 3 | 0
Death (General disorders) | 1 | 1
Dysphagia (General disorders) | 0 | 1
Gastrointestinal (Gastrointestinal disorders) | 4 | 0
Infection - Other (Infections and infestations) | 0 | 1
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 13 | 5
Neurological (Nervous system disorders) | 0 | 2
Other (General disorders) | 1 | 1
Pain - Back and/or Lower Extremities (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain - Upper Extremities (Musculoskeletal and connective tissue disorders) | 0 | 1
Psychological (Psychiatric disorders) | 1 | 0
Surgery - Adjacent Level (Surgical and medical procedures) | 4 | 2
Surgery - Index Level (Surgical and medical procedures) | 6 | 14
Surgery - Lumbar Level (Surgical and medical procedures) | 6 | 5
Surgery - Other Cervical (Surgical and medical procedures) | 0 | 1
Surgery - Thoracic Level (Surgical and medical procedures) | 1 | 0
Trauma (Injury, poisoning and procedural complications) | 0 | 1
Urogenital (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than .5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SECURE-C Cervical Artificial Disc (N=236) | ASSURE Cervical Plate and an Allograft Interbody Spacer (N=144)
Cancer (General disorders) | 2 | 0
Cardiovascular (Cardiac disorders) | 3 | 1
Carpal Tunnel Syndrome (CTS) (General disorders) | 6 | 5
Cerebrovascular (Vascular disorders) | 1 | 2
Compressive Peripheral Neuropathy (Non-CTS) (Nervous system disorders) | 4 | 0
Dysesthesia - Lower Extremities (Nervous system disorders) | 2 | 1
Dysesthesia - Other (Nervous system disorders) | 2 | 3
Dysesthesia - Upper Extremities (Nervous system disorders) | 20 | 15
Dysphagia (General disorders) | 6 | 7
Dysphonia (General disorders) | 1 | 2
Gastrointestinal (Gastrointestinal disorders) | 2 | 1
Headache (General disorders) | 8 | 11
Infection - Other (Infections and infestations) | 3 | 2
Infection - Superficial Wound (Infections and infestations) | 0 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 17 | 4
Neurological (Nervous system disorders) | 3 | 2
Other (General disorders) | 10 | 3
Pain - Back and/or Lower Extremities (General disorders) | 34 | 23
Pain - Neck (General disorders) | 50 | 41
Pain - Neck and Upper Extremities (General disorders) | 26 | 28
Pain - Neck and Upper Extremities with Dysesthesia (General disorders) | 1 | 3
Pain - Neck with Dysesthesia (General disorders) | 2 | 4
Pain - Other (General disorders) | 2 | 1
Pain - Upper Extremities (General disorders) | 32 | 23
Pain - Upper Extremities with Dysesthesia (General disorders) | 5 | 2
Psychological (Psychiatric disorders) | 0 | 1
Trauma (Injury, poisoning and procedural complications) | 30 | 16
Weakness (General disorders) | 3 | 1
Wound Issue (Skin and subcutaneous tissue disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
To prevent premature disclosure of information, Investigators agree not to present, publish, or disclose study results or information about the Investigational Device without the express written consent of Sponsor.